CLINICAL TRIAL: NCT04396704
Title: A Single Centre, Non-interventional, Retrospective Study to Assess Treatment Outcomes of abobotulinumtoxinA and onabotulinumtoxinA Treatments in Real Life Practice in Toxin-naïve Adult Patients With Limb Spasticity.
Brief Title: A Study to Assess Treatment Outcomes of abobotulinumtoxinA and onabotulinumtoxinA Treatments in Real Life Practice in Toxin-naïve Adult Patients With Limb Spasticity.
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: F-GB-52120-268
Record Dates: First submitted 2020-05-05; First posted 2020-05-20 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Spasticity Related to Any Cause Except Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Botox: all eligible subjects, in a reverse consecutive order, initiated on onaBoNT-A from 01 March 2015 to 29 May 2017.
- Dysport: all subjects meeting inclusion/exclusion criteria and initiated on aboBoNT-A from 30 May 2017 to 30 March 2019.

SUMMARY:
The aim of the study is to describe treatment outcomes of abobotulinumtoxinA (aboBoNT-A) and onabotulinumtoxinA (onaBoNT-A) treatments, after one injection of either treatment, in toxin-naïve adult patients with upper and/or lower limb spasticity at a single National Health Service (NHS) centre in the United Kingdom (UK).

ELIGIBILITY:
Inclusion Criteria :

* Patient diagnosed with spasticity related to any cause except cerebral palsy.
* Patient initiated on treatment with either onaBoNT-A or aboBoNT-A during the study enrolment periods.
* Patient is an adult aged ≥18 years old at the time of the first BoNT-A injection for spasticity
* Patient has not received treatment with any type of BoNT-A 6 months prior to initiation of onaBoNT-A or aboBoNT-A. For patients with multiple courses of BoNT-A, separated by a gap of 6 months, only the first course will be evaluated in this study.
* Patient is being treated at Haywood Hospital at index date and during follow-up for up to 24 weeks post-index date, with medical records available for review.

Exclusion Criteria :

* Patient is participating in an interventional clinical trial of an investigational medicinal product for the treatment of spasticity at index date and/or during follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult subjects with Upper Limb Spasticity and/or Lower Limb Spasticity complying with all inclusion and exclusion criteria during the study enrolment period will be included in this study. This study is retrospective and non-interventional, and as such, subjects will have been treated in accordance with usual medical practice during the study period. No additional assessments or tests will be required.
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Average Goal Attainment Scale (GAS T) score 6 weeks | 6 weeks
  GAS, a method that evaluates the attainment of priority goals that are of importance to the patient and has been previously used for the management of patients with limb spasticity. Rating is performed for each domain from -3 "worse than at start" to +2 "much more than expected: clear improvement".
Average Goal Attainment Scale (GAS T) score 12 weeks | 12 weeks
  GAS, a method that evaluates the attainment of priority goals that are of importance to the patient and has been previously used for the management of patients with limb spasticity. Rating is performed for each domain from -3 "worse than at start" to +2 "much more than expected: clear improvement".
Proportion of patients who achieve GAS-T score ≥0 for impairment/ symptoms goal | 12 weeks
Proportion of patients who exceed GAS-T score ≥1 for impairment/ symptoms goal | 6 weeks
Proportion of patients who exceed GAS-T score ≥1 for impairment/ symptoms goal | 12 weeks
Proportion of patients who achieve GAS-T score ≥0 for impairment/ symptoms goal | 6 weeks

SECONDARY OUTCOMES:
Average total dose | Day 0 (first BoNT-A injection) and from baseline up to 24 weeks (reinjection)
Average dose per limb and per type of muscle injected | Day 0 (first BoNT-A injection) and from baseline up to 24 weeks (reinjection)
Distribution of vials used | Day 0 (first BoNT-A injection) and from baseline up to 24 weeks (reinjection)
  If Dysport® 300U / 500U, if Botox® 50U / 100U / 200U
Distribution of localisation methods | Day 0 (first BoNT-A injection) and from baseline up to 24 weeks (reinjection)
  Ultrasound, electrostimulation, palpation, electromyography
Distribution of limb and type of muscles injected | Day 0 (first BoNT-A injection) and from baseline up to 24 weeks (reinjection)
  Upper limb: shoulder girdle, shoulder, arm, forearm, hand; lower limb: hip, thigh, leg and foot
Proportion of patients who require re-injection between aboBoNT-A and onaBoNT-A | Week 6 and week 12 (re-injection)
Quality of Life (QoL) | From baseline up to 12 weeks
  The EQ-5D-VAS is used to evaluate patients' quality of life. EQ-5D-VAS is one component of the EQ-5D-5L, a generic, preference-based measure of health-related quality of life. The questions are answered based on how the subject is feeling "today".
Average number of unscheduled visits | From baseline up to end of the study (up to 24 weeks)
Proportion of patients with ≥1 unscheduled visit | From baseline up to end of the study (up to 24 weeks)
Proportion of patients with at least "the same", or at least "better" satisfaction with their treatment as measured using a Likert scale | From baseline up to 12 weeks
  A Likert scale is used to record patient's satisfaction with his/her progress, and the patient's "best response" (since index date) and "response now" (at the time of the review) on a five-category scale: From "Much worse" to "Much better"

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- North Staffordshire Rehabilitation Centre. Midlands Partnership NHS Foundation Trust., Stafford, United Kingdom